CLINICAL TRIAL: NCT02940353
Title: The TREFOIL Concept: A Clinical Investigation in the Mandible on 3 Implants With a Fixed Prefabricated Framework
Brief Title: The TREFOIL Concept 5 Year Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-188
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2022-09

CONDITIONS: Edentulous or Failing Dentition Mandible
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Trefoil concept (Other): Treatment
  Interventions: Device: TREFOIL concept

INTERVENTIONS:
Device: TREFOIL concept

SUMMARY:
Prospective, single cohort, multi-center study evaluating the TREFOIL concept for the treatment of edentulous or patients with failing mandibular dentition over 5 years. 90 patients (15 per centre) will be included. The subject population is at least 18 years old, in need of an implant restored full prosthesis providing sufficient bone in the interforaminal where a fixed restoration on three implants is regarded as an appropriate treatment solution. The components are TREFOIL treatment concept (implants and framework).

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent from the subject.
* The subject is at least 18 years of age (passed cessation of growth) and not older than 80 years.
* The subject is in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems.
* The subject fulfills the prerequisite that a harmonic, stable occlusal relationship can be achieved with opposing natural teeth resp. fixed or removable opposing dentition (tooth or implant based) or soft tissue born denture.
* The subject is willing and able to comply with all study related procedures (such as exercising oral hygiene and attending all follow-up procedures).
* The subject is compliant with good oral hygiene.
* The subject has an edentulous mandible or failing mandibular dentition providing sufficient bone in the interforaminal where a fixed restoration on three (3) implants is regarded as an appropriate treatment solution.
* The subject has an osseous architecture enough to receive three implants with a length of at least 11.5 mm and a diameter of 5 mm in the interforaminal (e.g. jaw volume B, C or D; inter foramina distance at least 20 mm; buccal/lingual width at least 6-7 mm, vertical height after leveling bone sufficient to receive an implant of at least 11.5 mm length).
* The subject has a jaw curvature that fits to the prefabricated framework design.
* Implants will be placed in healed or extraction sites (clinical stability has to be ensured).
* The implant sites are free from infection and extraction remnants.
* The subjects as well as the implant sites fulfill the criteria for early loading.

Smokers that have reduced their consumption may be included after a certain test phase (e.g. test phase for reduction from 2 to 1 packages of cigarettes should be at least 6 months).

Class II inter-jaw relation patients are not an exclusion criteria per se. Based on the individual judgment of the clinician those patients may be treated.

Subject inclusion criteria at time of surgery

* After bone leveling sufficient mandible bone volume in the interforaminal present for three (3) implants with a length of at least 11.5 mm and a diameter of 5 mm.
* After bone leveling the jaw curvature does fit to the prefabricated framework.
* The implant sites are free from infection and extraction remnants.
* The subject as well as the implant sites fulfill the criteria for early loading.

Exclusion Criteria:

* The subject is not able to give her/his informed consent of participating.
* Health conditions, which do not permit the surgical (including anesthesia) or restorative procedure.
* Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or history.
* Any disorders in the planned implant area such as previous tumors, chronic bone disease or previous irradiation.
* Alcohol or drug abuse as noted in subject records or in subject history.
* Smoking of more than 1 package of cigarettes per day (> 20 cigarettes or equivalent).
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake or A1c level above 8%.
* Bisphosphonate therapy - based on individual judgment of the clinician (if intravenously administered or too high oral doses recently before surgery and during follow-up period).
* Pathologic occlusion, e.g. severe bruxism or other destructive habits.
* Lack of opposing dentition or unstable occlusion.
* Ongoing infections, endodontic or periodontal problems in opposing teeth or implants.
* Subject shows an unacceptable oral hygiene.
* Subject has allergic or adverse reactions to the restorative material.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-04; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Cumulative survival rates for the implants | 5 years

CONTACTS AND LOCATIONS:
Locations (5):
- Dr. Higuchi &Skinner, Spokane, Washington, United States
- Branemark Centre, Perth, Western Australia, Australia
- Clinica Rosenberg, Santiago, Santiago de Chile, Chile
- University of Verona, Verona, Italy
- Instituto Davó, Hospital Medimar Internacional, Alicante, Spain